CLINICAL TRIAL: NCT01319877
Title: A Multi-center Observational Study of Bevacizumab Plus 5-FU Based Chemotherapy as First Line and Second Line Treatment for Chinese Patients With Metastatic Colorectal Cancer (ML25391)
Brief Title: An Observational Study of Bevacizumab in Combination With 5-FU-Based Chemotherapy in Chinese Participants With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25391
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- First Line Treatment: Participants received bevacizumab in combination with 5-FU based chemotherapy as a first line therapy.
- Second Line Treatment: Participants received bevacizumab in combination with 5-FU based chemotherapy as a second line therapy.

SUMMARY:
This observational study will evaluate the safety and efficacy of Bevacizumab in combination with 5-Fluorouracil based chemotherapy as first-line and second-line therapy in Chinese participants with metastatic colorectal cancer. Data will be collected from each participant for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese participants, >/= 18 years of age
* Histologically confirmed and previously untreated metastatic colorectal cancer
* Initiated on treatment with Bevacizumab (in combination with 5-FU based chemotherapy) according to locally approved Bevacizumab China package insert
* Documented participant with medical records

Exclusion Criteria:

* Recent history of serious hemorrhage or hemoptysis of >/= 1/2 teaspoon of red blood
* Proteinuria at baseline (>/=2 grams / 24 hours)
* Major surgical procedure within 28 days prior to study treatment start, not fully healed wounds
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic colorectal cancer receiving first-line therapy with Bevacizumab in combination with 5-FU-based chemotherapy
Sampling Method: Probability Sample
Enrollment: 609 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- China (15):
  - Beijing
  - Changzhou
  - Chengdu
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Harbin
  - Jinan
  - Nanjing
  - Nanning
  - Shanghai
  - Shenyang
  - Wuhan
  - Xi'an
  - Xiamen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three enrolled participants received third-line therapy and were not included in the evaluable population.
Period: Overall Study
Arm/Group | First Line Treatment | Second Line Treatment
Started | 453 | 153
Completed | 345 | 108
Not Completed | 108 | 45
Not completed — Lost to Follow-up | 100 | 37
Not completed — Physician Decision | 2 | 0
Not completed — Disease Progression | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Reason Not Specified | 4 | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set and efficacy analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | First Line Treatment | Second Line Treatment | Total
Number analyzed (Participants) | 453 | 153 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.9) | 54.5 (11.9) | 55.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 53 | 236
  Male | 270 | 100 | 370
Region of Enrollment [Number; unit: participants]
  China | 453 | 153 | 606

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant after administration of a pharmaceutical product and which did not necessarily have a causal relationship with this treatment.
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 76.4 | 68.0

2. Primary Outcome: Percentage of Participants With Serious Adverse Events
Description: A Serious Adverse Event (SAE) was any untoward medical occurrence that at any dose was fatal, required inpatient hospitalization or prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant, or required intervention to prevent one or other of the outcomes listed above.
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 4.9 | 4.6

3. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 9.1 | 5.9

4. Primary Outcome: Percentage of Participants With Bevacizumab-Related Adverse Events
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 54.5 | 45.8

5. Primary Outcome: Percentage of Participants With Bevacizumab-related Serious Adverse Events
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 3.1 | 2.0

6. Secondary Outcome: Percentage of Participants Achieving an Overall Response
Description: Overall response was defined as complete response (CR) or partial response (PR) confirmed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, all non-target lesions, and no new lesions. PR: At least a 30% decrease in the sum of the diameters of target lesions, no progression in non-target lesions, and no new lesions.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 21.0 [17.3 to 25.0] | 10.5 [6.1 to 16.4]

7. Secondary Outcome: Progression-free Survival
Description: Progression-free-survival (PFS) was defined as the time from the date when the participant signed the informed consent form to the time of first documented disease progression or death, whichever occurred first.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
months | 9.1 [8.2 to 10.0] | 8.1 [6.0 to 11.0]

8. Secondary Outcome: One-year Progression-free Survival Rate
Description: One year progression-free survival rate was defined as the percentage of participants who were free of progression or death from the date when the participant signed the informed consent form to one year.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 34.2 [26.8 to 41.7] | 29.9 [18.6 to 42.1]

9. Secondary Outcome: One-year Survival Rate
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants | 68.7 [62.7 to 74.0] | 69.1 [59.1 to 77.2]

10. Secondary Outcome: Percentage of Participants Achieving an Overall Response Per Kirsten Rat Sarcoma Viral (KRAS) Oncogene Subgroup
Description: Overall response was defined as complete response (CR) or partial response (PR) confirmed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, all non-target lesions, and no new lesions. PR: At least a 30% decrease in the sum of the diameters of target lesions, no progression in non-target lesions, and no new lesions. Results are reported per participants' Kirsten Rat Sarcoma Viral (KRAS) oncogene subgroup.
Time Frame: 36 months
Population: Participants with known KRAS status were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants
  Wild-type | 18.6 [9.7 to 30.9] | 10.3 [2.2 to 27.4]
  Mutant-type | 10.7 [5.0 to 19.4] | 4.8 [0.1 to 23.8]

11. Secondary Outcome: One-year Progression-free Survival Rate Per KRAS Subgroup
Description: One year progression-free survival rate was defined as the percentage of participants who were free of progression or death from the date when the participant signed the informed consent form to one year. Results are reported per participants' Kirsten Rat Sarcoma Viral (KRAS) oncogene subgroup.
Time Frame: 1 year
Population: Participants with known KRAS status were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants
  Wild-type | 45.2 [22.6 to 65.4] | 31.3 [8.8 to 57.3]
  Mutant-type | 19.5 [7.5 to 35.6] | 0 [0 to 0]

12. Secondary Outcome: One-year Survival Rate by the KRAS Subgroup
Time Frame: 1 year
Population: Participants with known KRAS status were evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants
  Wild-type | 81.0 [64.7 to 90.3] | 69.1 [43.4 to 84.9]
  Mutant-type | 57.9 [42.7 to 70.4] | 33.9 [8.4 to 62.2]

13. Secondary Outcome: Percentage of Participants Achieving an Overall Response by the Chemotherapy Regimen Subgroup
Description: Overall response was defined as complete response (CR) or partial response (PR) confirmed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, all non-target lesions, and no new lesions. PR: At least a 30% decrease in the sum of the diameters of target lesions, no progression in non-target lesions, and no new lesions. Results are reported per participants' chemotherapy regimen subgroup.
Time Frame: Up to 36 Months
Population: Participants with known prior chemotherapy regimens were evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants
  FOLFOX | 25.7 [19.4 to 32.9] | 15.2 [5.1 to 31.9]
  IFL | 18.5 [12.9 to 25.4] | 10.9 [5.3 to 19.1]
  XELIRI | 45.5 [16.7 to 76.6] | 14.3 [0.4 to 57.9]
  XELOX | 32.1 [19.9 to 46.3] | 0 [0 to 41.0]
  Others | 5.8 [1.2 to 15.9] | 7.1 [0.2 to 33.9]

14. Secondary Outcome: One-year Progression-free Survival Rate Per Chemotherapy Regimen Subgroup
Description: One year progression-free survival rate was defined as the percentage of participants who were free of progression or death from the date when the participant signed the informed consent form to one year. Results are reported per participants' chemotherapy regimen subgroup.
Time Frame: 1 year
Population: Participants with known prior chemotherapy regimens were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants
  FOLFOX | 38.9 [28.1 to 49.5] | 38.1 [16.0 to 60.1]
  IFL | 29.1 [16.9 to 42.4] | 32.2 [16.5 to 49.1]
  XELIRI | 13.3 [0.8 to 43.3] | 20.0 [0.8 to 58.2]
  XELOX | 44.9 [17.1 to 69.6] | 20.8 [0.9 to 59.5]
  Others | 19.5 [3.6 to 45.0] | 16.7 [0.8 to 51.7]

15. Secondary Outcome: One-year Survival Rate by the Chemotherapy Regimen Subgroup
Time Frame: 1 year
Population: Participants with known prior chemotherapy regimens were evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 453 | 153
percentage of participants
  FOLFOX | 66.6 [56.8 to 74.7] | 71.6 [47.0 to 86.2]
  IFL | 70.8 [60.6 to 78.8] | 71.4 [58.2 to 81.0]
  XELIRI | 66.7 [27.2 to 88.1] | 20.8 [0.9 to 59.5]
  XELOX | 75.2 [56.1 to 86.9] | 0 [0 to 0]
  Others | 64.7 [38.4 to 82.0] | 60.0 [25.3 to 82.7]

16. Secondary Outcome: Quality of Life: European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 Questionnaire
Description: Quality of life was assessed at baseline and every three months after treatment by the EORTC QLQ-C30 questionnaire. The possible score range was 0 to 100, with a higher score indicating better functioning.
Time Frame: Up to 36 Months
Population: Evaluable participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 248 | 67
score on a scale
  Baseline (n=248,67) | 63.68 (18.020) | 65.67 (14.103)
  Visit 2 (n=159,44) | 62.89 (15.875) | 64.96 (17.105)
  Visit 3 (n=80,21) | 59.79 (18.073) | 56.35 (19.168)
  Visit 4 (n=50,12) | 54.83 (22.718) | 61.11 (14.360)
  Visit 5 (n=26,9) | 57.05 (15.758) | 62.96 (16.724)
  Visit 6 (n=15,5) | 57.22 (14.389) | 73.33 (16.030)
  Visit 7 (n=11,4) | 56.82 (16.168) | 72.92 (15.773)
  Visit 8 (n=7,3) | 60.72 (14.205) | 66.67 (8.335)
  Visit 9 (n=4,1) | 45.83 (15.960) | 66.67 (NA) — Not calculable, due to single data point.
  Visit 10 (n=1,0) | 50.00 (NA) — Not calculable, due to single data point. | NA (NA) — Not calculable, due to no participants for this data point.

ADVERSE EVENTS:
Time Frame: Up to 36 months
Groups:
- First and Second Line Treatment: The participants from the first line and second line treatments were combined for the adverse event analysis.
Arm/Group | First and Second Line Treatment
Serious Adverse Events (participants affected / at risk) | 29/606
Other Adverse Events (participants affected / at risk) | 450/606
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First and Second Line Treatment (N=606)
Enteritis (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Infection (Infections and infestations) | 2
Bacteremia (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Deep vein thrombosis (Vascular disorders) | 4
Myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 2
Neutrophil count decreased (Investigations) | 2
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Ureteric fistula (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | First and Second Line Treatment (N=606)
Nausea (Gastrointestinal disorders) | 108
Vomiting (Gastrointestinal disorders) | 93
Diarrhea (Gastrointestinal disorders) | 65
Constipation (Gastrointestinal disorders) | 31
White blood cell count decreased (Investigations) | 130
Neutrophil count decreased (Investigations) | 100
Platelet count decreased (Investigations) | 39
Alanine aminotransferase increased (Investigations) | 37
Aspartate aminotransferase increased (Investigations) | 36
Pyrexia (General disorders) | 58
Fatigue (General disorders) | 52
Bone marrow failure (Blood and lymphatic system disorders) | 73
Decreased appetite (Metabolism and nutrition disorders) | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.